CLINICAL TRIAL: NCT02763657
Title: Neural Development of Deductive Reasoning: an fMRI Study of Relational and Categorical Reasoning in Children
Brief Title: Neural Development of Deductive Reasoning
Acronym: NEUREAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012.767
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: fMRI; reasoning; development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain activity during reasoning (Experimental)
  Interventions: Other: fMRI scanning

INTERVENTIONS:
Other: fMRI scanning — All participants are scanned while evaluating linear-order and set-inclusion reasoning problems

SUMMARY:
Children's understanding of linear-order (e.g., Dan is taller than Lisa, Lisa is taller than Jess) and set-inclusion (i.e., All tulips are flowers, All flowers are plants) relationships is critical for the acquisition of deductive reasoning, that is, the ability to reach logically valid conclusions from given premises. Behavioral and neuroimaging studies in adults suggest processing differences between these relations: While arguments that involve linear-orders may be preferentially associated with spatial processing, arguments that involve set-inclusions may be preferentially associated with verbal processing. In this study, we use functional magnetic resonance imaging to investigate how and when these processing differences appear in children from 8 to 14.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Affiliated to the French social security
* Whose parents gave informed consent

Exclusion Criteria:

* Neurological disorders
* Psychiatric disorders
* Birth complications requiring admission into neonatal intensive care unit
* Medication affecting central nervous system processing
* Significant hearing impairment
* Uncorrected visual impairment
* Non-native English speaker
* Contraindications for MRI

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Identification of brain regions engaged in linear-order and set-inclusion reasoning | 30 days
  Brain activity measured using fMRI

SECONDARY OUTCOMES:
Degree of overlap between brain regions involved in linear-order and set-inclusion reasoning | 30 days
  Degree of overlap in brain activity measured using fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon/bron, France

IPD SHARING:
Plan to Share IPD: No